CLINICAL TRIAL: NCT04743713
Title: Turkish Cross-cultural Adaptation, Validation and the Reliability of UWRI (University of Wisconsin Running Injury and Recovery Index)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Elif Turgut, Assistant Professor (asst. prof.), Hacettepe University
Other Study IDs: GO 21/27
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Running Related Injuries
Keywords: validity; reliability; PRO; Patient Outcome Report; Turkish; Adaptation; Running; Injury
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: UWRI-Tr — Questionnaire

SUMMARY:
The purpose is to perform a scientific study on TURKISH cross-cultural adaptation, validation and the reliability of UWRI

DETAILED DESCRIPTION:
The primary aim of this study is to perform Turkish cross-cultural adaptation, validation and the reliability of UWRI in runners. The secondary aim of this study is investigating injury rate and types among runners.

ELIGIBILITY:
Inclusion Criteria:

* 14-45 years old female or male
* Participating in running as amateur, recreational, competitional or professional runner
* Being a short, mid, or long distance runner
* Being native Turkish speaker
* Agreed to participate in the research

Exclusion Criteria:

* If there is no surgical history related to running injury in the last 12 months
* If have chronic metabolic disease
* Paralympic athletes
* Pregnant and breastfeeding

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Runners
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-02-10 (Estimated); Primary Completion 2022-01-16 (Estimated); Study Completion 2022-01-16 (Estimated)

PRIMARY OUTCOMES:
Validity and reliability | 5-7 days
  pearson's correlation 2 tailed analysis; >0,60 good, 0,31-0,59 medium, <0,30 bad

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No